CLINICAL TRIAL: NCT02271100
Title: Assessment of the Use of Ultrasound for Epidural Catheter Placement and Comparison With Palpation Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014P000267
Record Dates: First submitted 2014-10-17; First posted 2014-10-22 (Estimated); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: randomized blinded comparison of two methods to identify landmarks for a procedure
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- palpation guidance (Placebo Comparator): placement of spinal or combined spinal epidural needle using palpation to guide entry position
  Interventions: Device: palpation guidance
- ultrasound guidance (Active Comparator): placement of spinal or combined spinal epidural using ultrasound to guide entry position
  Interventions: Device: ultrasound guidance

INTERVENTIONS:
Device: ultrasound guidance — use of ultrasound for entry position estimation
  Arms: ultrasound guidance
Device: palpation guidance — use of palpation for position estimation
  Arms: palpation guidance

SUMMARY:
This study is intended to determine whether ultrasound imaging can improve the ability to place a spinal or epidural needle in obstetric anesthesia. By evaluating the use of ultrasound for the placement of epidural catheters the investigators hope to answer two questions:

1. How does the traditional technique based on palpation compare to one using ultrasound to place an epidural catheter? 2. Does ultrasound reduce one potential risk in epidural placement?

DETAILED DESCRIPTION:
This study contains two phases:

1. A prospective, randomized, blinded comparison of ultrasound imaging versus palpation for epidural catheter insertion in laboring women.
2. A prospective, single cohort, blinded trial to assess whether ultrasound imaging provides a reliable placement below the L3 vertebra.

The initial phase of the investigation will be a randomized comparison of ultrasound versus palpation. Patients will be enrolled in early labor and will be randomized to have their epidural placed with either technique. The technique will be chosen by computer-generated randomization list maintained in opaque sequentially numbered envelopes. Description of the placement technique is below. The primary outcome will be the number of epidural catheters inserted above the intended insertion site. The investigators will also assess the total time required for epidural catheter placement, number of attempts for successful insertion, effectiveness of the epidural catheter for labor pain control.

Following completion of enrollment of the first phase, the second phase of the investigation will enroll patients only into the single-cohort ultrasound arm. The study will use the same methodology as the initial phase, but without randomization due to a single cohort. The primary outcome will be the absolute number of epidural catheters inserted above the L3 vertebral body. The investigators will also assess the effectiveness of the ultrasound markings for guiding placement.

Procedure placement technique After written, informed consent, and standard patient preparation, the epidural catheter will be placed with the patient in the sitting position by a junior resident. In the ultrasound arm, the patient will be first imaged using an appropriate probe, and the identified ultrasound landmarks marked on the skin. The skin will be prepped in the usual fashion, and the needle will be inserted at the identified site and direction determined by ultrasound. In the palpation arm, the skin will be prepped and the needle will be inserted using palpation-identified landmarks to guide the needle. All catheters will be intended to be placed at the L4-L5 interspace as the primary attempt. The L3-L4 interspace will be used as a secondary attempt.

Assessment of final position After insertion of the epidural catheter and administration of the pain relief medication, patients in both groups will be examined by a blinded observer using ultrasound to determine the catheter insertion site and the likely insertion interspace.

If, however, the investigators discover that the use of ultrasound for placement of the epidural catheter may present greater risk than previously anticipated to the pregnant woman or fetus, then the investigators will stop the study after phase 1 and not proceed with phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ASA I or II parturient
* Will be receiving neuraxial placement for labor, having been consented for the procedure

Exclusion Criteria:

* ASA III or IV
* Unable to participate in the study due to severe pain
* Contraindications to neuraxial analgesia
* Previous spinal surgery in the lumbar or sacral area (L1 through Sacrum)
* BMI greater than 37
* Height less than 60 inches
* Significant scoliosis

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Placement below L3 vertebra | immediate
  Percentage of catheters placed below the target location

SECONDARY OUTCOMES:
Time to placement | immediate
  Minutes from start of procedure to the end of the procedure
Success of the epidural catheter placement | immediate
  Relief of labor pain defined by verbal pain score less than 4 after administration of medication

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Hess, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Isreal Deaconess Medical Center, Boston, Massachusetts, United States